CLINICAL TRIAL: NCT04758286
Title: Protocol for Anesthesia for Emergency Surgery
Brief Title: Anesthetic & Surgical Protocol for Emergency Surgeries During the Era of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Adel F. Alkholy, Professor of Medical Biochemistry, Benha University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RC2-2-2021
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: COVID-19; Anesthesia; Surgery; Outcomes
MeSH Terms: conditions — COVID-19 | interventions — Anesthesia, Spinal; Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: All patients presenting with surgical emergency
Who Masked: Outcomes Assessor
Masking Description: An anesthetist who was not in charge for application of the protocol is responsible for assessing the intraoperative findings and another anesthetist was responsible for assessing the postoperative findings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successful outcome (Active Comparator): It will include the anesthetic and operative data and the incidence of intraoperative or postoperative complication
  Interventions: Procedure: Emergency surgical procedures
- Complicated outcome (Active Comparator): It will include the anesthetic and operative data and the incidence of intraoperative or postoperative complication
  Interventions: Procedure: Emergency surgical procedures

INTERVENTIONS:
Procedure: Emergency surgical procedures — COVID-19 patients who had presented to the Emergency Department were evaluated for their emergency surgical conditions and were managed appropriately
  Other Names: Spinal anesthesia; Epidural anesthesia; Total intravenous anesthesia

SUMMARY:
A protocol applied during anesthesia and surgical interventions for patients with emergency surgical conditions during the era of COVID-19 disease

DETAILED DESCRIPTION:
All COVID-19 patients who were admitted to emergency departments presenting with emergency surgical conditions were evaluated for assurance of having COVID-19 disease. Then, the appropriate anesthetic procedure was applied and the appropriate surgical intervention was performed.

ELIGIBILITY:
Inclusion Criteria:

* Assured diagnosis of COVID-19 by RT-PCR

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Up to two days
  This questionnaire was designed to assess the satisfaction of the anesthetist in-charge and the surgeon by the applied protocol to manage COVID-19 patients

SECONDARY OUTCOMES:
Physiologic assessment | Up to one day
  estimation of systolic and diastolic blood pressures of patients during and after surgery
Surgical follow-up | Up to 10 days
  Postoperative assessment of wounds and drainage tube, if any, and to determine the success of the procedure or the development of complications

CONTACTS AND LOCATIONS:
Overall Officials: Adel Alkholy, Prof, Principal Investigator — Faculty of medicine, Banha University, Egypt
Locations (1):
- Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol may be shared
Supporting Information: Study Protocol
Time Frame: after publishing
Access Criteria: email